CLINICAL TRIAL: NCT03068442
Title: Amyloid Deposition and Preexisting Vulnerable Carotid Plaque Features Predicting Cognitive Improvement After Surgery
Brief Title: The Role of Large Artery Plaque Imaging Features in Predicting Inflammation and Cognition
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scott Mcnally (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Scott Mcnally, Assistant Professor, Department of Radiology, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17SDG33460420
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Impairment; Carotid Artery Plaque; Inflammation
Keywords: Carotid artery; MRI; PET; Intraplaque hemorrhage
MeSH Terms: conditions — Cognitive Dysfunction; Carotid Stenosis; Inflammation | interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: This is a diagnostic-interventional cohort study in patients undergoing carotid endarterectomy for atherosclerotic disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carotid atherosclerosis group (Experimental): This group includes all enrolled subjects (those with carotid disease and plans to undergo surgery).
  Interventions: Drug: Imaging with flutemetamol F 18 PET/CT

INTERVENTIONS:
Drug: Imaging with flutemetamol F 18 PET/CT — All subjects will undergo diagnostic imaging as the intervention. This imaging will be with flutemetamol F 18 PET/CT

SUMMARY:
The invesigators propose a clinical study on patients undergoing carotid surgery (endarterectomy). The invesigators will determine carotid artery imaging features associated with (1) vessel wall inflammation, (2) downstream brain inflammation, and (3) cognitive benefit from surgery. This project will uncover links between inflamed carotid plaque and downstream brain inflammation. The invesigators will also determine carotid plaque imaging features predicting cognitive benefit from carotid surgery.

DETAILED DESCRIPTION:
This research is directed at a major stroke source, the carotid artery, a major vessel that supplies blood to the brain. It has long been known that carotid narrowing is an important stroke risk factor. However, many patients with narrow carotids do not have strokes, and many patients with seemingly normal carotids have strokes. MRI research now suggests that the carotid wall itself is the stroke source. Using carotid MRI, clinicians can identify previously invisible markers of unstable carotid plaque, including carotid wall bleeds (intraplaque hemorrhage). The working hypothesis is that patients with these unstable carotid plaques may have higher inflammation in both their carotid arteries and brain. This inflammation has been implicated in other diseases, including dementia.

Carotid wall bleeds can easily be seen with carotid MRI, but are often invisible on ultrasound and CT scans. By using MRI, the invesigators have found that this silent killer is an important stroke risk factor even without carotid narrowing. Now that imaging can detect carotid wall bleeds, where do the bleeds come from? Recent research points to inflammation within the carotid wall. The invesigators plan to use histology to detect this inflammation in the vessel wall. Another question is, does inflammation in the carotid wall lead to inflammation in the brain? Using PET scans, the invesigators plan to determine whether inflammation in the brain is linked to carotid disease. Lastly, the invesigators hope to find out if carotid wall inflammation contributes to memory loss and if surgery is beneficial in these patients.

The invesigators hope to detect this inflammation in the vessel wall and brain before patients develop stroke, memory loss and dementia. This will be of huge benefit not only in the detection of diseases, but would also allow clinicians to monitor treatment effect on both carotid disease and brain inflammation. The invesigators also hope to use these tools to detect early treatment response. This research will accelerate the pace of future clinical trials to bring important new medications to patients sooner.

ELIGIBILITY:
Inclusion Criteria:

• Patients ≥18 years old and plans for carotid endarterectomy.

Exclusion Criteria:

* Patients with carotid occlusion will be excluded, due to one carotid contributing to both right and left brain blood supply.
* Other known sources of cardioembolism, including atrial fibrillation, mechanical heart valve, left atrial or ventricular thrombus or intracardiac mass, endocarditis, EF <30%
* Known stroke mimics including multiple sclerosis or brain tumor
* MRI contraindications per ACR guidelines, including patients with pacemakers, renal failure with eGFR<30 ml/min/1.73m2, and contrast allergy
* [18F]Flutemetamol contraindications per manufacturer guidelines, including patients with prior reactions
* Known stage IV malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Carotid intraplaque hemorrhage correlation with carotid plaque inflammation on immunohistochemistry. | baseline
  Carotid plaque inflammation will be calculated with quantitative immunohistochemistry and correlated with intraplaque hemorrhage while controlling for confounders.
Carotid MRI-detected intraplaque hemorrhage and prediction of brain inflammation on PET/CT. | baseline
  Outcome 2. The primary outcome, brain inflammation will be compared in carotid intraplaque hemorrhage positive and negative sides, controlling for confounders including stenosis and perfusion.
Preoperative MRI-detected carotid intraplaque hemorrhage and prediction of cognitive improvement after endarterectomy. | Change from baseline at 3 month followup
  Outcome 3. The primary outcome, difference in cognitive score will be compared in carotid intraplaque hemorrhage positive and negative patients, controlling for stenosis, perfusion and ischemic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S McNally, MD, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All data will be made freely and publicly available on ClinicalTrials.gov within 12 months of the end of the funding period (and any no-cost extension).
  1. Carotid intraplaque hemorrhage
  2. Carotid plaque inflammation on histology
  3. Age, stroke status, male sex, smoking and vitamin D level
  4. Statin, antiplatelet, or antihypertensive use
  5. Ipsilateral brain inflammation measured by PET
  6. Carotid stenosis and perfusion parameters
  7. Cognitive score